CLINICAL TRIAL: NCT04934475
Title: MInimal Residual Disease Adapted Strategy: Frontline Therapy for Patients Eligible for Autologous Stem Cell Transplantation Less Than 66 Years; a Prospective Study
Brief Title: MInimal Residual Disease Adapted Strategy
Acronym: MIDAS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Intergroupe Francophone du Myelome (Network)
Collaborators: Amgen (Industry); Sanofi (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: IFM2020-02; 2020-005216-21 (EudraCT Number)
Record Dates: First submitted 2021-05-11; First posted 2021-06-22 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-11

CONDITIONS: Multiple Myeloma
Keywords: Younger patients; First line of treatment; Autograft; Isa-KRD
MeSH Terms: conditions — Multiple Myeloma | interventions — isatuximab; carfilzomib; Lenalidomide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: All patients will receive ISa-KRD treatment for induction. Depending on MRD status, patients will be randomized :
  MRD Standard-risk post induction MRD <10-5,(1:1 Randomization):
  Arm A: 6 additional cycles of Isa-KRD Arm B: ASCT followed by 2 cycles of Isa-KRD MRD High-risk (post induction MRD >10-5) (1:1 Randomization) Arm C: ASCT followed by 2 cycles of Isa-KRD Arm D: tandem ASCT
  Maintenance:
  In arms A/B, patients will receive commercial Lenalidomide, for 3 years. In arms C/D, patients will receive Iberdomide and Isatuximab for 3 years. Treatment allocation A/B to patients: randomization stratified per center according to LP score.
  Treatment allocation C/D to patients: randomization stratified per center according to LP score.
  For each randomization, primary analysis will evaluate MRD (NGS, 10-6 threshold) after all subjects have completed the post-consolidation response evaluation or have been discontinued from study treatment by this timepoint
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- MRD Standard-risk patients (post induction MRD <10-5, MRD SR) (1:1 Randomization) : Arm A (Experimental): Arm A: consolidation with 6 additional cycles of Isa-KRD (cycles 7 to 12; 28-day cycle; Isa-KRD = Isatuximab Carfilzomib Lenalidomide Dexamethasone):
  * Isatuximab: 10 mg/kg I.V. on days 1 and 15 (cycles 7 to 12)
  * Carfilzomib: 56 mg/m2 I.V on days 1, 8 and 15 (cycles 7 to 12)
  * Lenalidomide: 25 mg per day orally from days 1 to 21
  * Dexamethasone: 40 mg orally on day 1, 8, 15, 22
  Interventions: Drug: Isatuximab
- MRD Standard-risk patients (post induction MRD <10-5, MRD SR) (1:1 Randomization): Arm B (Experimental): Arm B: consolidation with ASCT followed by 2 cycles of Isa-KRD (cycles 7 and 8; Isa-KRD = Isatuximab Carfilzomib Lenalidomide Dexamethasone; 28-day cycle) Melphalan 200 mg/m2 followed by autologous stem cell transplantation (please refer to section 6.3.2)
  * Isatuximab: 10 mg/kg I.V. on days 1 and 15 (cycles 7 to 8)
  * Carfilzomib: 56 mg/m2 I.V on days on days 1, 8 and 15 (cycles 7 to 8)
  * Lenalidomide: 25 mg per day orally from days 1 to 21
  * Dexamethasone: 40 mg orally on days 1, 8, 15, 22 (cycles 7 to 8)
  Interventions: Drug: Isatuximab; Procedure: ASCT
- MRD High-risk patients (post induction MRD >10-5, MRD HR) (1:1 Randomization): Arm C (Experimental): Arm C: ASCT followed by 2 cycles of Isa-KRD (cycles 7 and 8; Isa-KRD = Isatuximab Carfilzomib Lenalidomide Dexamethasone; 28-day cycle) Melphalan 200 mg/m2 followed by autologous stem cell transplantation.
  * Isatuximab: 10 mg/kg I.V. on days 1 and 15 (cycles 7 to 8)
  * Carfilzomib: 56 mg/m2 I.V on days on days 1, 8 and 15 (cycle 7 to 8)
  * Lenalidomide: 25 mg per day orally from day 1 to day 21
  * Dexamethasone: 40 mg orally on days 1, 8, 15, 22 (cycle 7 to 8)
  Interventions: Drug: Isatuximab; Procedure: ASCT
- MRD High-risk patients (post induction MRD >10-5, MRD HR) (1:1 Randomization): Arm D (Experimental): Tandem ASCT Melphalan 200 mg/m2 followed by autologous stem cell transplantation.
  Interventions: Procedure: ASCT

INTERVENTIONS:
Drug: Isatuximab — Treatment with Isa-KRD during induction and consolidation , with Lenalidomide (Revlimid) or Iberdomide + Isatuximab during maintenance phase
  Other Names: Carfilzomib; Revlimid; Dexamethasone
  Arms: MRD High-risk patients (post induction MRD >10-5, MRD HR) (1:1 Randomization): Arm C; MRD Standard-risk patients (post induction MRD <10-5, MRD SR) (1:1 Randomization) : Arm A; MRD Standard-risk patients (post induction MRD <10-5, MRD SR) (1:1 Randomization): Arm B
Procedure: ASCT — ASCT for ams B, C and D during consolidation
  Arms: MRD High-risk patients (post induction MRD >10-5, MRD HR) (1:1 Randomization): Arm C; MRD High-risk patients (post induction MRD >10-5, MRD HR) (1:1 Randomization): Arm D; MRD Standard-risk patients (post induction MRD <10-5, MRD SR) (1:1 Randomization): Arm B

SUMMARY:
IFM 2020-02 will enroll patients eligible for ASCT less than 66 years. All patients will receive induction based on 6 cycles (28-day) of KRD-Isatuximab (Isa-KRD), in order to achieve deep responses and high MRD negativity rates. Patients will be classified at diagnosis according to cytogenetics (standard vs high-risk cytogenetics defined by the LP score including 17p deletion, t(4;14), del(1p32), gain 1q, trisomy 21 and trisomy 5).

DETAILED DESCRIPTION:
According to international guidelines, outside clinical trials, frontline autologous stem cell transplantation (ASCT) is the standard of care for fit patients less than 71 years of age, who are newly diagnosed with multiple myeloma.

Triplet combinations are now the backbone of induction therapy prior to ASCT. KRD (Carfilzomib, Lenalidomide, Dexamethasone) is potentially the more active regimen.

Quadruplet combinations are under evaluation. The prospective phase 3 CASSIOPEIA trial conducted by the IFM and HOVON cooperative groups investigated the outcome of transplant-eligible patients treated with VTD (Bortezomib, Thalidomide, Dexamethasone) +/- Daratumumab administered both before (induction, 4 cycles) and after (consolidation, 2 cycles) single ASCT prepared by Melphalan 200 mg/m2.5 The addition of Daratumumab to VTD during induction induced significantly higher response rates, but also higher minimal residual disease (MRD) - negativity rates. The high response rates achieved after induction (MRD negativity rates at 10-5 by 8-color flow cytometry 35% (188/543) in the VTD-Dara arm vs 23% (125/542) after 4 cycles of VTD in the intent-to-treat population), but also after consolidation and before maintenance (MRD negativity rates at 10-5 by 8-color flow cytometry 63% in the VTD-Dara arm vs 43% in the VTD in the intent-to-treat population), translated into a significant improvement in progression-free-survival (PFS) in the Daratumumab arm of the study: 18-month PFS 93% vs 85% before maintenance, HR 0.47 (0.33-0.67), p < 0.0001. Cassiopeia is the first study showing a correlation between MRD negativity after induction (before ASCT) and PFS benefit, in the setting of quadruplet combination induction. Based on these results, VTD + daratumumab was recently approved by the FDA and EMA.

KRD has also been combined with Daratumumab in several phase 2 trials. Early results indicate that this quadruplet combination might potentially be the most effective regimen prior to ASCT in terms of response and MRD-negativity rates. Carfilzomib was administered intravenously weekly, on days 1, 8 and 15 of 28 day-cycles at the dose of 56 mg/m². Based on 70 patients, the MRD-negativity rate after four cycles of KRD-Daratumumab was 39% at a detection level of 10-5 by next generation sequencing (NGS). The weekly KRD-Daratumumab regimen was associated with low toxicity, and stem cell harvest was adequate. The rate of MRD negativity in 42 patients further improved after single ASCT, to 67% and 43% at a detection level of 10-5 and of 10-6 by NGS, respectively. Due to the short 7.9 months median follow-up time at the time of presentation, no PFS data were presented. At ASCO 2020, Weisel et al reported the results of induction based on 6 cycles of KRD plus Isatuximab, in patients with high-risk cytogenetics.8 In this interim analysis on the first 46 patients eligible for ASCT with high-risk disease, the overall response rate was 100%, including 60% MRD negativity at 10-5 by NGS after induction and before ASCT. No death on study was reported. No data are yet available regarding MRD negativity rates after ASCT or PFS. At ASH 2019, Landgren et al. reported the results of eight weekly KRD-Daratumumab cycles without ASCT in a small phase 2 study on 41 patients after a short median follow-up time of 8.6 months.

On the same intent-to-treat basis, MRD-negativity rate at a detection level of 10-5 by NGS was 61% and 65% in patients after six and eight cycles, respectively, including a very good partial response (VGPR) rate or better of 85% after 8 cycles and an overall response rate (ORR) of 100%. No death on study was seen. At the time of the report, no patient with MRD-negative disease had progressed. Despite the short follow-up time, based on the high rate of MRD-negativity and the 0% relapse rate achieved so far with this quadruplet combination, the authors of this small phase 2 series now propose to systematically delay ASCT in patients with standard-risk disease. This provocative recommendation requires validation in a phase 3 randomized trial comparing frontline versus delayed ASCT in patients with MRD-negative disease after induction.

Patients MRD positive after quadruplet induction are at higher risk of disease progression. For patients with high-risk (HR) disease, tandem ASCT has been proposed in order to improve PFS and overall survival (OS). In an integrated analysis of four phase III studies independently conducted by HOVON/GMMG, IFM, PETHEMA/GEM and GIMEMA European cooperative groups, in the era of Bortezomib-based induction regimens, double ASCT significantly improved PFS and OS in HR patients.

In the EMN02/HO95 study, in centers with a policy of double ASCT, patients were assigned to receive VMP (Bortezomib, Melphalan, Prednisone), single ASCT (ASCT-1) or two planned ASCTs (ASCT-2) to prospectively compare ASCT-1 with ASCT-2. Patients who received ASCT-2 had a prolonged PFS compared to those who received ASCT-1. Importantly, ASCT-2 overcame the adverse prognosis conferred by high-risk cytogenetics. In the same study, OS from the first randomization was significantly prolonged with ASCT-2 as compared with ASCT-1, a benefit also seen in subgroups of patients with adverse prognosis, including those with R-ISS stage II+III and high-risk cytogenetics. To date, no prospective trial has compared single vs tandem ASCT in HR patients in the era of quadruplet induction combinations.

After ASCT, a systematic maintenance is recommended by International Guidelines. Lenalidomide is approved in this setting, and proposed until progression. Other agents or combinations are under evaluation for maintenance, such as Ixazomib, Elotuzumab, Daratumumab or Isatuximab. Iberdomide is a next generation cereblon targeting agent, with antitumor and immunostimulatory activities in Lenalidomide- and Pomalidomide-resistant multiple myeloma. This oral agent, which could be the ideal agent for maintenance therapy, is currently tested after ASCT. Phase 2 and 3 randomized studies are currently investigating the combination of Lenalidomide with anti-CD38 monoclonal antibodies as maintenance therapy after autologous stem cell transplant. We assume that a fixed duration of maintenance using Iberdomide and Isatuximab will induce a high-rate of sustained MRD negativity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, 18 years of age or older, younger than 66 years (< 66 years)
2. Voluntary written informed consent must be given before performance of any study-related procedure not part of normal medical care, with the understanding that the subject may withdraw consent at any time without prejudice to future medical care.
3. Subject must have documented multiple myeloma satisfying the CRAB and measurable disease as defined by:

   1. Monoclonal plasma cells in the bone marrow ≥ 10% or presence of a biopsy proven plasmacytoma AND any one or more of the following myeloma defining events:

      * Hypercalcemia: serum calcium > 0.25 mmol/L (> 1 mg/dL) higher than ULN or > 2.75 mmol/L (> 11 mg/dL)
      * Renal insufficiency: creatinine clearance < 40mL/min or serum creatinine > 177 μmol/L (> 2 mg/dL)
      * Anemia: hemoglobin > 2 g/dL below the lower limit of normal or hemoglobin < 10 g/dL
      * Bone lesions: one or more osteolytic lesions on skeletal radiography, CT or PET-CT
      * Clonal bone marrow plasma cell percentage ≥ 60%
      * Involved: uninvolved serum free light chain ratio ≥ 100
      * Superior 1 focal lesion on MRI studies
   2. Measurable disease as defined by the following:

      * M-component ≥ 5g/L, and/or urine M-component ≥ 200 mg/24h and/or serum FLC ≥ 100 mg/L
4. Newly diagnosed subjects eligible for high dose therapy and autologous stem cell transplantation
5. Karnofsky performance status score ≥ 50% (eastern cooperative oncology group performance status ECOG score ≤ 2)
6. Subject must have pretreatment clinical laboratory values meeting the following criteria during the Screening Phase (Lab tests should be repeated if done more than 15 days before C1D1):

   1. Hemoglobin ≥ 7.5 g/dL (≥ 5mmol/L). Prior red blood cell [RBC] transfusion or recombinant human erythropoietin use is permitted;
   2. Absolute neutrophil count (ANC) ≥ 1.0 Giga/L (GCSF use is permitted);
   3. ASAT ≤ 3 x ULN;
   4. ALAT ≤ 3 x ULN;
   5. Total bilirubin ≤ 3 x ULN (except in subjects with congenital bilirubinemia, such as Gilbert syndrome, direct bilirubin ≤ 1.5 x ULN);
   6. Calculated creatinine clearance ≥ 40 mL/min/1.73 m²;
   7. Corrected serum calcium ≤ 14 mg/dL (< 3.5 mmol/L); or free ionized calcium ≤6.5 mg/dL (≤ 1.6 mmol/L);
   8. Platelet count ≥ 50 Giga/L for subjects in whom < 50% of bone marrow nucleated cells are plasma cells; otherwise platelet count > 50 Giga/L (transfusions are not permitted to achieve this minimum platelet count).
7. Women of childbearing potential must have a negative serum or urine pregnancy test within 10 to 14 days prior to therapy and repeated within 24 hours before starting study drug. They must commit to continued abstinence from heterosexual intercourse or begin 2 acceptable methods of birth control (One highly effective method and one additional effective method) used at the same time, beginning at least 4 weeks before initiation of Lenalidomide treatment and continuing for at least 30 days after the last dose of Lenalidomide, Iberdomide and 5 months after last dose of Isatuximab. Women must also agree to notify pregnancy during the study.
8. Men must agree to not father a child and agree to use a latex condom during therapy and during dose interruptions and for at least 90 days after the last dose of study drug including Lenalidomide and Iberdomide and 5 months after last dose of Isatuximab, even if they have had a successful vasectomy, if their partner is of childbearing potential. Patient must also refrain from donating sperm during this period.

Exclusion Criteria:

1. Subjects must not have been treated previously with any systemic therapy for multiple myeloma. Prior treatment with corticosteroids or radiation therapy does not disqualify the subject (the maximum dose of corticosteroids should not exceed the equivalent of 160 mg of dexamethasone in a 2-week period). Two weeks must have elapsed since the date of the last radiotherapy treatment. Enrolment of subjects who require concurrent radiotherapy (which must be localized in its field size) should be deferred until the radiotherapy is completed and 2 weeks have elapsed since the last date of therapy.
2. Subject has a diagnosis of primary amyloidosis, monoclonal gammopathy of undetermined significance, smoldering multiple myeloma, or solitary plasmacytoma.
3. Subject has a diagnosis of Waldenström's macroglobulinemia, or other conditions in which IgM M-protein is present in the absence of a clonal plasma cell infiltration with lytic bone lesions.
4. Subject has had plasmapheresis within 14 days of C1D1.
5. Subject is exhibiting clinical signs of meningeal involvement of multiple myeloma.
6. Myocardial infarction within 4 months prior to enrolment according to NYHA Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities
7. Uncontrolled hypertension
8. Subjects with a history of moderate or severe persistent asthma within the past 2 years, or with uncontrolled asthma of any classification at the time of screening (Note that subjects who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed in the study).
9. Intolerance to hydration due to pre-existing pulmonary or cardiac impairment.
10. Subject has plasma cell leukemia (according to WHO criterion: ≥ 20% of cells in the peripheral blood with an absolute plasma cell count of more than 2 × 109/L) or POEMS syndrome (polyneuropathy, organomegaly, endocrinopathy, monoclonal protein, and skin changes).
11. Any clinically significant, uncontrolled medical conditions that, in the Investigator's opinion, would expose the patient to excessive risk or may interfere with compliance or interpretation of the study results.
12. Systemic treatment with strong inhibitors of CYP1A2 (fluvoxamine, enoxacin), strong inhibitors of CYP3A (clarithromycin, telithromycin, itraconazole, voriconazole, ketoconazole, nefazodone, posaconazole) or strong CYP3A inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of Ginkgo biloba or St. John's wort within 14 days before the first dose of study treatment.
13. Known intolerance to steroid therapy, mannitol, pregelatinized starch, odium stearyl fumarate, histidine (as base and hydrochloride salt), arginine hydrochloride, poloxamer 188, sucrose or any of the other components of study intervention that are not amenable to premedication with steroids and H2 blockers or would prohibit further treatment with these agents.
14. History of allergy to any of the study medications, their analogues, or excipients in the various formulations
15. Subject has had major surgery within 2 weeks before study inclusion (informed consent signature) or will not have fully recovered from surgery, or has surgery planned during the time the subject is expected to participate in the study. Kyphoplasty or Vertebroplasty are not considered major surgery.
16. Clinically relevant active infection or serious co-morbid medical conditions
17. Prior malignancy except adequately treated basal cell or squamous cell skin cancer, in situ cervical, breast or prostate cancer free of disease since 5 years.
18. Female subject who is pregnant or breast-feeding
19. Serious medical or psychiatric illness likely to interfere with participation in study
20. Uncontrolled diabetes mellitus
21. Known HIV infection; Known active hepatitis A, B or C viral infection
22. Uncontrolled or active HBV infection: Patients with positive HBsAg and/or HBV DNA

    Of note:
    * Patient can be eligible if anti-HBc IgG positive (with or without positive anti-HBs) but HBsAg and HBV DNA are negative.
    * If anti-HBV therapy in relation with prior infection was started before initiation of IMP, the anti-HBV therapy and monitoring should continue throughout the study treatment period.
    * Patients with negative HBsAg and positive HBV DNA observed during screening period will be evaluated by a specialist for start of anti-viral treatment: study treatment could be proposed if HBV DNA becomes negative and all the other study criteria are still met.
23. Active HCV infection: positive HCV RNA and negative anti-HCV

    Of note:
    * Patients with antiviral therapy for HCV started before initiation of IMP and positive HCV antibodies are eligible. The antiviral therapy for HCV should continue throughout the treatment period until seroconversion.
    * Patients with positive anti-HCV and undetectable HCV RNA without antiviral therapy for HCV are eligible.
24. Active systemic infection and severe infections requiring treatment with a parenteral administration of antibiotics.
25. Incidence of gastrointestinal disease that may significantly alter the absorption of oral drugs
26. Subjects unable or unwilling to undergo antithrombotic prophylactic treatment
27. Person under guardianship, trusteeship or deprived of freedom by a judicial or administrative decision

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 791 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2028-09-30 (Estimated)

PRIMARY OUTCOMES:
Negative MRD rate | Time Frame: change from post induction baseline MRD at end of consolidation phase (6 months)
  For both parts of the trial (A vs B and C vs D), the primary comparison of the 2 strategies will be made with respect to negative MRD rate (10-6 NGS) before maintenance using the chi square test in the ITT population.
  The observed MRD negative rate will be provided along with its 2-sided 95% Confidence interval (CI). Treatment effect will be described by an Odds Ratio, along with its 2-sided 95% confidence interval, by fitting a logistic regression model adjusted on stratification variables (with high risk cytogenetics and MRD negative rate (10-5 NGS) after induction as fixed effects and center as random effects for A vs B comparison, and high risk cytogenetics as fixed effects and center as random effects for C vs D comparison). In case of missing MRD, data will be imputed as positive in all arms.
  Sensitivity analyses will be performed using best-worst and worst-best case to check for robustness of the results.
Negative MRD rate | change from post induction baseline MRD at 1 years
  For both parts of the trial (A vs B and C vs D), the primary comparison of the 2 strategies will be made with respect to negative MRD rate (10-6 NGS) before maintenance using the chi square test in the ITT population.
  The observed MRD negative rate will be provided along with its 2-sided 95% Confidence interval (CI). Treatment effect will be described by an Odds Ratio, along with its 2-sided 95% confidence interval, by fitting a logistic regression model adjusted on stratification variables (with high risk cytogenetics and MRD negative rate (10-5 NGS) after induction as fixed effects and center as random effects for A vs B comparison, and high risk cytogenetics as fixed effects and center as random effects for C vs D comparison). In case of missing MRD, data will be imputed as positive in all arms.
  Sensitivity analyses will be performed using best-worst and worst-best case to check for robustness of the results.
Negative MRD rate | change from post induction baseline MRD at 2 years
  For both parts of the trial (A vs B and C vs D), the primary comparison of the 2 strategies will be made with respect to negative MRD rate (10-6 NGS) before maintenance using the chi square test in the ITT population.
  The observed MRD negative rate will be provided along with its 2-sided 95% Confidence interval (CI). Treatment effect will be described by an Odds Ratio, along with its 2-sided 95% confidence interval, by fitting a logistic regression model adjusted on stratification variables (with high risk cytogenetics and MRD negative rate (10-5 NGS) after induction as fixed effects and center as random effects for A vs B comparison, and high risk cytogenetics as fixed effects and center as random effects for C vs D comparison). In case of missing MRD, data will be imputed as positive in all arms.
  Sensitivity analyses will be performed using best-worst and worst-best case to check for robustness of the results.
Negative MRD rate | change from post induction baseline MRD at 3 years
  For both parts of the trial (A vs B and C vs D), the primary comparison of the 2 strategies will be made with respect to negative MRD rate (10-6 NGS) before maintenance using the chi square test in the ITT population.
  The observed MRD negative rate will be provided along with its 2-sided 95% Confidence interval (CI). Treatment effect will be described by an Odds Ratio, along with its 2-sided 95% confidence interval, by fitting a logistic regression model adjusted on stratification variables (with high risk cytogenetics and MRD negative rate (10-5 NGS) after induction as fixed effects and center as random effects for A vs B comparison, and high risk cytogenetics as fixed effects and center as random effects for C vs D comparison). In case of missing MRD, data will be imputed as positive in all arms.
  Sensitivity analyses will be performed using best-worst and worst-best case to check for robustness of the results.

SECONDARY OUTCOMES:
Sustained MRD rate | change from post induction baseline MRD at end of consolidation phase (6 months)
  Sustained MRD rate at after consolidation phase ( 6 months) than year 1, 2, 3 post consolidation phase will be analyzed similarly to the primary endpoint
Sustained MRD rate | change from post induction baseline MRD at 1 years
  Sustained MRD rate at after consolidation phase ( 6 months) than year 1, 2, 3 post consolidation phase will be analyzed similarly to the primary endpoint
Sustained MRD rate | change from post induction baseline MRD at 2 years
  Sustained MRD rate at after consolidation phase ( 6 months) than year 1, 2, 3 post consolidation phase will be analyzed similarly to the primary endpoint
Sustained MRD rate | change from post induction baseline MRD at 3 years
  Sustained MRD rate at after consolidation phase ( 6 months) than year 1, 2, 3 post consolidation phase will be analyzed similarly to the primary endpoint
Overall Survival (OS) | through study completion, an average of 8 year
  For Overall Survival (OS), the distribution of OS since randomization will be estimated using Kaplan Meier method. The comparison of the 2 arms will be made by log-rank test. Treatment effect will be described by Hazard Ratio and its 2-sided 95% confidence intervals will be estimated using a Cox regression model adjusted on stratification variables (with high risk cytogenetics and MRD negative rate (10-5 NGS) after induction as fixed effects and center as random effects for A vs B comparison, and high risk cytogenetics as fixed effects and center as random effects for C vs D comparison).
Progression Free Survival (PFS) | through study completion, an average of 8 year
  Progression Free Survival, defined as time from randomization to either progression or death will be analyzed similarly to OS
Safety analyses | until 30 days post last dose of protocol treatment
  rate of adverse events that occured during treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Moreau, Professor, Principal Investigator — Nantes University Hospital
Locations (73):
- Belgium (6):
  - Institut Jules Bordet, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - Grand Hôpital de Charleroi - Site de Notre-Dame, Charleroi
  - Hôpital Jolimont, Haine-Saint-Paul
  - CHU de Liège, Liège
  - CHU UCL Namur (Site Godinne), Yvoir
- France (66):
  - CHU Amiens Sud, Amiens
  - CHRU-Hôpital du Bocage, Angers
  - Centre Hospitalier d'Argenteuil Victor Dupouy, Argenteuil
  - Centre Hospitalier H.Duffaut, Avignon
  - Centre hospitalier de la Côte Basque, Bayonne
  - Hôpital Jean Minjoz, Besançon
  - Centre Hospitalier Simone Veil, Blois
  - Hôpital Avicenne, Bobigny
  - Polyclinique Bordeaux Nord Acquitaine, Bordeaux
  - CHRU Hôpital Haut Lévêque - Centre François Magendie, Bordeaux Pessac
  - Hôpital de Fleyriat, Bourg-en-Bresse
  - CHRU Brest - Hôpital A. Morvan, Brest
  - CHU Caen - Côte de Nacre, Caen
  - CH René Dubos, Cergy-Pontoise
  - Centre Hospitalier William Morey, Chalon-sur-Saône
  - CH Chambéry, Chambéry
  - Hôpital d'Instruction des Armées Percy, Clamart
  - Chu Estaing, Clermont-Ferrand
  - Centre Hospitalier Sud Francilien, Corbeil-Essonnes
  - CHU Henri Mondor, Créteil
  - CHU Dijon Hôpital d'enfants, Dijon
  - Centre Hospitalier Général, Dunkirk
  - CHRU Hôpital A. Michallon, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - CHV André Mignot - Université de Versailles, Le Chesnay
  - CH de Chartres - Hôpital Louis Pasteur, Le Coudray
  - Hôpital Jacques Monod, Le Havre
  - Centre Hospitalier, Le Mans
  - CHRU Hôpital Claude Huriez, Lille
  - GH de l'Institut Catholique Saint Vincent, Lille
  - Centre Hospitalier Universitaire (CHU) de Limoges, Limoges
  - Hôpital du Scorff, Lorient
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - CH Meaux, Meaux
  - Hôpital de Mercy (CHR Metz-Thionville), Metz
  - Hopital Saint Eloi - CHU Montpellier, Montpellier
  - Hôpital E. Muller, Mulhouse
  - CHRU Hôtel Dieu, Nantes
  - Clinique de l'Archet, Nice
  - CHU Carémeau, Nîmes
  - CH La Source, Orléans
  - CHU Hôpital Saint Antoine, Paris
  - Hôpital Cochin, Paris
  - Hôpital Necker, Paris
  - Hôpital Saint Louis, Paris
  - Institut Curie, Paris
  - La Pitié- Salpetrière, Paris
  - CH Saint Jean, Perpignan
  - Centre Hospitalier de Perigueux, Périgueux
  - Hospices Civils de Lyon - Hôpital Lyon Sud, Pierre-Bénite Lyon
  - CHU Poitiers - Pôle régional de Cancérologie, Poitiers
  - Ch Annecy Genevois, Pringy
  - Centre Hospitalier Intercommunal de Cornouaille, Quimper
  - Hôpital Robert Debré, Reims
  - CHRU Hôpital de Pontchaillou, Rennes
  - Centre Henri Becquerel, Rouen
  - Centre Hospitalier Yves Le Foll, Saint-Brieuc
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin
  - Hôpitaux Universitaires de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - Pôle IUCT Oncopole CHU, Toulouse
  - CHRU Hôpital Bretonneau, Tours
  - CHRU Hôpitaux de Brabois, Vandœuvre-lès-Nancy
  - CHBA, Vannes
  - Gustave Roussy, Villejuif
- CHU de La Réunion site Sud, Saint-Pierre, Reunion

REFERENCES:
- [Derived] Perrot A, Lambert J, Hulin C, Pieragostini A, Karlin L, Arnulf B, Rey P, Garderet L, Macro M, Escoffre-Barbe M, Gay J, Chalopin T, Gounot R, Schiano JM, Mohty M, Leleu X, Manier S, Mariette C, Chaleteix C, Braun T, De Prijck B, Avet-Loiseau H, Mary JY, Corre J, Moreau P, Touzeau C; MIDAS Study Group. Measurable Residual Disease-Guided Therapy in Newly Diagnosed Myeloma. N Engl J Med. 2025 Jul 31;393(5):425-437. doi: 10.1056/NEJMoa2505133. Epub 2025 Jun 3. PMID 40459097
- [Derived] Perrot A, Touzeau C, Lambert J, Hulin C, Caillot D, Karlin L, Arnulf B, Rey P, Garderet L, Macro M, Escoffre Barbe M, Gay J, Chalopin T, Gounot R, Schiano JM, Tiab M, Mohty M, Kuhnowski F, Fontan J, Manier S, Orsini-Piocelle F, Vincent L, Rigaudeau S, Leleu X, Hebraud B, Flet L, Malfuson JV, Jacquet C, Chaoui D, Meuleman N, Abarah W, Montes L, Benramdane R, Sonntag C, Zerazhi H, Danu A, Allangba O, Dib M, Roussel M, Cereja S, Depaus J, Branche N, Demarquette H, Richez V, Cherel B, Frenzel L, Vekemans MC, Bigot N, Avet-Loiseau H, Corre J, Moreau P. Isatuximab, carfilzomib, lenalidomide, and dexamethasone induction in newly diagnosed myeloma: analysis of the MIDAS trial. Blood. 2025 Jul 3;146(1):52-61. doi: 10.1182/blood.2024026230. PMID 39841461
- [Derived] Mohan M, Gundarlapalli S, Szabo A, Yarlagadda N, Kakadia S, Konda M, Jillella A, Fnu A, Ogunsesan Y, Yarlagadda L, Thalambedu N, Munawar H, Graziutti M, Al Hadidi S, Alapat D, Thanendrarajan S, Zangari M, van Rhee F, Schinke C. Tandem autologous stem cell transplantation in patients with persistent bone marrow minimal residual disease after first transplantation in multiple myeloma. Am J Hematol. 2022 Jun 1;97(6):E195-E198. doi: 10.1002/ajh.26530. Epub 2022 Mar 21. No abstract available. PMID 35285981